CLINICAL TRIAL: NCT04455932
Title: HCC Surveillance: Comparison of Abbreviated Non-contrast MRI and Ultrasound Surveillance in Cirrhotic Patients With Suboptimal Ultrasound Visualisation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concord Repatriation General Hospital (Other)
Responsible Party: Principal Investigator, Dr Jessica Yang, Principal Investigator, Concord Repatriation General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019/PID15472
Record Dates: First submitted 2020-06-27; First posted 2020-07-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma; HCC
Keywords: Ultrasound; MRI; HCC; Hepatocellular carcinoma; aMRI; NC-aMRI; Screening; Surveillance
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCC surveillance with US and aNC-MRI (Experimental)
  Interventions: Diagnostic Test: Abbreviated non-contrast MRI of the liver; Diagnostic Test: Ultrasound surveillance; Diagnostic Test: Multiphase contrast-enhanced liver MRI

INTERVENTIONS:
Diagnostic Test: Abbreviated non-contrast MRI of the liver — every 6 months
  Other Names: aNC-MRI
Diagnostic Test: Ultrasound surveillance — every 6 months
  Other Names: US surveillance
Diagnostic Test: Multiphase contrast-enhanced liver MRI — screening
  Other Names: Multiphase liver MRI

SUMMARY:
All international guidelines recommend 6-monthly ultrasound surveillance for patients at risk for liver cancer (hepatocellular carcinoma or HCC), such as patients with cirrhosis. The aim of surveillance is to detect HCC at an early stage when it is still potentially curable. Currently only 4 out of 10 HCCs are detected at the early stage.

Ultrasound surveillance for HCC has a wide ranging sensitivity, dependent on many factors such as operator experience, patient body habitus and liver parenchymal heterogeneity due to chronic liver disease and cirrhosis. In a select group of patients, surveillance ultrasound can be suboptimal or near non-diagnostic.

Currently no guideline offers an alternative surveillance tool for patients who have suboptimal surveillance ultrasounds.

DETAILED DESCRIPTION:
The investigators plan to conduct a prospective study to examine the diagnostic performance of abbreviated non-contrast MRI (aNC-MRI) versus ultrasound, in a select group of cirrhotic patients with poor ultrasound visualisation.

ELIGIBILITY:
Inclusion criteria

* Patients with cirrhosis (all causes of cirrhosis, except obscure causes such as vascular or congenital fibrosis) AND reduced visualisation of their liver on ultrasound (vB and vC).
* The criteria of cirrhosis can be obtained with any of the following methods:

  1. Histologically by liver biopsy
  2. Past signs of decompensated liver disease such as ascites, encephalopathy, varices or bacterial peritonitis
  3. Clinically suspicion of cirrhosis PLUS one of the following:

     1. Radiological evidence of morphologic changes of the liver and evidence of portal hypertension on US, CT or MRI examinations, including the identification of hepatic surface nodularity, splenomegaly, portal collaterals, varices and ascites
     2. Fibroscan (transient elastography) median liver stiffness >12.5 kPa, the Fibroscan must be performed by an experienced technician and interpreted by the hepatologist
     3. Platelet count <100 (x10^9/L) with no alternative cause
* Absence of previous history or current suspicion of HCC - Absence of HCC is defined by liver US, multiphase CT or contrast-enhanced MRI within 6 months prior to surveillance
* Patient is able to comply with scheduled visits, evaluation plans and other study procedures in the opinion of the investigator
* Patient is willing to provide written informed consent

Exclusion criteria

* Contraindications to MRI scan (defibrillator, pacemaker, metallic foreign body, severe claustrophobia etc.)
* Contraindications to gadolinium
* Age above 85 years old or younger than 20 years old
* Pregnancy or breast feeding
* Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrolment for the trial or could interfere with the completion of the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
HCC detection with US surveillance versus aNC-MRI surveillance | 3 or 5 years
  The detection of hepatic malignancy on the two modalities will be compared
  * Sensitivity, specificity, PPV and NPV of HCC detection with US surveillance vs aNC-MRI surveillance
  * Correlation with diagnostic imaging (multiphase CT or MRI) and/or histopathology as a reference standard
  For the diagnosis of HCC we will accept
  * Imaging diagnosis based on the Liver Imaging Reporting and Data System (LI-RADS)
  * Any pathological proof on biopsy or excision The HCC will then be staged based on the Barcelona clinic liver cancer (BCLC) staging system
  For the diagnosis of non-HCC hepatic malignancy we will accept
  * Imaging diagnosis based on the Liver Imaging Reporting and Data System (LI-RADS)
  * Any pathological proof on biopsy or excision

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yang, MBBS, Principal Investigator — Concord Repatriation General Hospital
Locations (10):
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- North Shore Hospital, Takapuna, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Son JH, Choi SH, Kim SY, Jang HY, Byun JH, Won HJ, Lee SJ, Lim YS. Validation of US Liver Imaging Reporting and Data System Version 2017 in Patients at High Risk for Hepatocellular Carcinoma. Radiology. 2019 Aug;292(2):390-397. doi: 10.1148/radiol.2019190035. Epub 2019 Jun 18. PMID 31210614
- [Result] Singal AG, Pillai A, Tiro J. Early detection, curative treatment, and survival rates for hepatocellular carcinoma surveillance in patients with cirrhosis: a meta-analysis. PLoS Med. 2014 Apr 1;11(4):e1001624. doi: 10.1371/journal.pmed.1001624. eCollection 2014 Apr. PMID 24691105
- [Result] Tzartzeva K, Obi J, Rich NE, Parikh ND, Marrero JA, Yopp A, Waljee AK, Singal AG. Surveillance Imaging and Alpha Fetoprotein for Early Detection of Hepatocellular Carcinoma in Patients With Cirrhosis: A Meta-analysis. Gastroenterology. 2018 May;154(6):1706-1718.e1. doi: 10.1053/j.gastro.2018.01.064. Epub 2018 Feb 6. PMID 29425931
- [Result] Hanna RF, Miloushev VZ, Tang A, Finklestone LA, Brejt SZ, Sandhu RS, Santillan CS, Wolfson T, Gamst A, Sirlin CB. Comparative 13-year meta-analysis of the sensitivity and positive predictive value of ultrasound, CT, and MRI for detecting hepatocellular carcinoma. Abdom Radiol (NY). 2016 Jan;41(1):71-90. doi: 10.1007/s00261-015-0592-8. PMID 26830614
- [Result] Colli A, Fraquelli M, Casazza G, Massironi S, Colucci A, Conte D, Duca P. Accuracy of ultrasonography, spiral CT, magnetic resonance, and alpha-fetoprotein in diagnosing hepatocellular carcinoma: a systematic review. Am J Gastroenterol. 2006 Mar;101(3):513-23. doi: 10.1111/j.1572-0241.2006.00467.x. PMID 16542288
- [Result] Chernyak V, Fowler KJ, Kamaya A, Kielar AZ, Elsayes KM, Bashir MR, Kono Y, Do RK, Mitchell DG, Singal AG, Tang A, Sirlin CB. Liver Imaging Reporting and Data System (LI-RADS) Version 2018: Imaging of Hepatocellular Carcinoma in At-Risk Patients. Radiology. 2018 Dec;289(3):816-830. doi: 10.1148/radiol.2018181494. Epub 2018 Sep 25. PMID 30251931
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] D'Avola D, Labgaa I, Villanueva A. Natural history of nonalcoholic steatohepatitis/nonalcoholic fatty liver disease-hepatocellular carcinoma: Magnitude of the problem from a hepatology clinic perspective. Clin Liver Dis (Hoboken). 2016 Oct 27;8(4):100-104. doi: 10.1002/cld.579. eCollection 2016 Oct. No abstract available. PMID 31041073
- [Result] Saunders D, Seidel D, Allison M, Lyratzopoulos G. Systematic review: the association between obesity and hepatocellular carcinoma - epidemiological evidence. Aliment Pharmacol Ther. 2010 May;31(10):1051-63. doi: 10.1111/j.1365-2036.2010.04271.x. Epub 2010 Feb 18. PMID 20175765
- [Result] Wang C, Wang X, Gong G, Ben Q, Qiu W, Chen Y, Li G, Wang L. Increased risk of hepatocellular carcinoma in patients with diabetes mellitus: a systematic review and meta-analysis of cohort studies. Int J Cancer. 2012 Apr 1;130(7):1639-48. doi: 10.1002/ijc.26165. Epub 2011 Jul 28. PMID 21544812
- [Result] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Result] Chitturi S, Wong VW, Chan WK, Wong GL, Wong SK, Sollano J, Ni YH, Liu CJ, Lin YC, Lesmana LA, Kim SU, Hashimoto E, Hamaguchi M, Goh KL, Fan J, Duseja A, Dan YY, Chawla Y, Farrell G, Chan HL. The Asia-Pacific Working Party on Non-alcoholic Fatty Liver Disease guidelines 2017-Part 2: Management and special groups. J Gastroenterol Hepatol. 2018 Jan;33(1):86-98. doi: 10.1111/jgh.13856. No abstract available. PMID 28692197
- [Result] Benson AB 3rd, D'Angelica MI, Abbott DE, Abrams TA, Alberts SR, Saenz DA, Are C, Brown DB, Chang DT, Covey AM, Hawkins W, Iyer R, Jacob R, Karachristos A, Kelley RK, Kim R, Palta M, Park JO, Sahai V, Schefter T, Schmidt C, Sicklick JK, Singh G, Sohal D, Stein S, Tian GG, Vauthey JN, Venook AP, Zhu AX, Hoffmann KG, Darlow S. NCCN Guidelines Insights: Hepatobiliary Cancers, Version 1.2017. J Natl Compr Canc Netw. 2017 May;15(5):563-573. doi: 10.6004/jnccn.2017.0059. PMID 28476736
- [Result] Burak KW, Sherman M. Hepatocellular carcinoma: Consensus, controversies and future directions. A report from the Canadian Association for the Study of the Liver Hepatocellular Carcinoma Meeting. Can J Gastroenterol Hepatol. 2015 May;29(4):178-84. doi: 10.1155/2015/824263. PMID 25965437
- [Result] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Result] Kokudo N, Hasegawa K, Akahane M, Igaki H, Izumi N, Ichida T, Uemoto S, Kaneko S, Kawasaki S, Ku Y, Kudo M, Kubo S, Takayama T, Tateishi R, Fukuda T, Matsui O, Matsuyama Y, Murakami T, Arii S, Okazaki M, Makuuchi M. Evidence-based Clinical Practice Guidelines for Hepatocellular Carcinoma: The Japan Society of Hepatology 2013 update (3rd JSH-HCC Guidelines). Hepatol Res. 2015 Jan;45(2). doi: 10.1111/hepr.12464. PMID 25625806
- [Result] Marrero JA, Ahn J, Rajender Reddy K; Americal College of Gastroenterology. ACG clinical guideline: the diagnosis and management of focal liver lesions. Am J Gastroenterol. 2014 Sep;109(9):1328-47; quiz 1348. doi: 10.1038/ajg.2014.213. Epub 2014 Aug 19. PMID 25135008
- [Result] Korean Liver Cancer Study Group (KLCSG); National Cancer Center, Korea (NCC). 2014 KLCSG-NCC Korea Practice Guideline for the Management of Hepatocellular Carcinoma. Gut Liver. 2015 May 23;9(3):267-317. doi: 10.5009/gnl14460. PMID 25918260
- [Result] Besa C, Lewis S, Pandharipande PV, Chhatwal J, Kamath A, Cooper N, Knight-Greenfield A, Babb JS, Boffetta P, Padron N, Sirlin CB, Taouli B. Hepatocellular carcinoma detection: diagnostic performance of a simulated abbreviated MRI protocol combining diffusion-weighted and T1-weighted imaging at the delayed phase post gadoxetic acid. Abdom Radiol (NY). 2017 Jan;42(1):179-190. doi: 10.1007/s00261-016-0841-5. PMID 27448609
- [Result] Tillman BG, Gorman JD, Hru JM, Lee MH, King MC, Sirlin CB, Marks RM. Diagnostic per-lesion performance of a simulated gadoxetate disodium-enhanced abbreviated MRI protocol for hepatocellular carcinoma screening. Clin Radiol. 2018 May;73(5):485-493. doi: 10.1016/j.crad.2017.11.013. Epub 2017 Dec 12. PMID 29246586
- [Result] Lee JY, Huo EJ, Weinstein S, Santos C, Monto A, Corvera CU, Yee J, Hope TA. Evaluation of an abbreviated screening MRI protocol for patients at risk for hepatocellular carcinoma. Abdom Radiol (NY). 2018 Jul;43(7):1627-1633. doi: 10.1007/s00261-017-1339-5. PMID 29018942
- [Result] Chan MV, McDonald SJ, Ong YY, Mastrocostas K, Ho E, Huo YR, Santhakumar C, Lee AU, Yang J. HCC screening: assessment of an abbreviated non-contrast MRI protocol. Eur Radiol Exp. 2019 Dec 18;3(1):49. doi: 10.1186/s41747-019-0126-1. PMID 31853685
- [Result] Park SH, Kim B, Kim SY, Shim YS, Kim JH, Huh J, Kim HJ, Kim KW, Lee SS. Abbreviated MRI with optional multiphasic CT as an alternative to full-sequence MRI: LI-RADS validation in a HCC-screening cohort. Eur Radiol. 2020 Apr;30(4):2302-2311. doi: 10.1007/s00330-019-06546-5. Epub 2019 Dec 19. PMID 31858203
- [Result] Lewis S, Kamath A, Chatterji M, Patel A, Shyknevsky I, Dyvorne HA, Kuehn B, Taouli B. Diffusion-weighted imaging of the liver in patients with chronic liver disease: comparison of monopolar and bipolar diffusion gradients for image quality and lesion detection. AJR Am J Roentgenol. 2015 Jan;204(1):59-68. doi: 10.2214/AJR.13.11695. PMID 25539238
- [Result] Whang S, Choi MH, Choi JI, Youn SY, Kim DH, Rha SE. Comparison of diagnostic performance of non-contrast MRI and abbreviated MRI using gadoxetic acid in initially diagnosed hepatocellular carcinoma patients: a simulation study of surveillance for hepatocellular carcinomas. Eur Radiol. 2020 Aug;30(8):4150-4163. doi: 10.1007/s00330-020-06754-4. Epub 2020 Mar 12. PMID 32166493
- [Result] Marrero JA, Kulik LM, Sirlin CB, Zhu AX, Finn RS, Abecassis MM, Roberts LR, Heimbach JK. Diagnosis, Staging, and Management of Hepatocellular Carcinoma: 2018 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2018 Aug;68(2):723-750. doi: 10.1002/hep.29913. No abstract available. PMID 29624699
- See also: US LIRADS CORE 2017 — https://www.acr.org/-/media/ACR/Files/RADS/LI-RADS/CEUS-LI-RADS-2017-Core.pdf?la=en%20n.d